CLINICAL TRIAL: NCT01317628
Title: Effects of Tobacco Smoke Exposure on Epigenetic Signatures and Immunotoxicological Reactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201009040R
Record Dates: First submitted 2011-03-08; First posted 2011-03-17 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: The Study Focused on Reducing Tobacco Smoke Exposure for Child.
Keywords: tobacco smoke, intervention program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Other): Both the parents and children will receive 8 times intervention program weekly in first session. The telephone counseling will reduce the child's tobacco smoke exposure every weekly in second session. The interventionist and child jointly select behavioral goals for reducing tobacco smoke exposure for the child to work toward. The goals will be formalized as a written smoke exposure reduction plan for any of four specific behaviors, as relevant to that family: (a) smoking cessation for the child, (b) making the child's primary home smoke-free, (c) making non-home locations smoke-free.
  Interventions: Behavioral: Tobacco smoke reduction trial intervention program

INTERVENTIONS:
Behavioral: Tobacco smoke reduction trial intervention program — Both the parents and children will receive 8 times intervention program weekly in first session. The telephone counseling will reduce the child's tobacco smoke exposure every weekly in second session. The interventionist and child jointly select behavioral goals for reducing tobacco smoke exposure for the child to work toward. The goals will be formalized as a written smoke exposure reduction plan for any of four specific behaviors, as relevant to that family: (a) smoking cessation for the child, (b) making the child's primary home smoke-free, (c) making non-home locations smoke-free.

SUMMARY:
Researchers have noted that active smoke exposure was possibly related to epigenetic mechanism,and may further influence reactive immunotoxicological reaction on human beings. Some studies have been reported that smoking reduction would decrease the prevalence of respiratory symptoms and urinary cotinine level, but the underlying epigenetic mechanism and the functional changes of immunotoxicological system were still unclear. We plan to examine the causal relationship between smoking reduction and alterations in epigenetic signatures/immunotoxicological reactions. Teenager Smoking Reduction Trial (TSRT) will be population-based trial among teenagers. Eligible teenagers will be recruited in Taipei City and urinary cotinine level will be used to monitor the exposure status of active smoking at baseline, 1-month and 3-month of the intervention process. We will assess the potential change in immunotoxicological markers, including Th1/Th2 cytokines and clinical immunological measurements, before and after the intervention program. Furthermore, whole-genome methylation and miRNA expression microarrays will be used to search candidate genes for teenager smoking exposure. We plan to develop a prediction model for immunotoxicological reaction by utilizing epigenetic signature data from microRNA expression and DNA methylation profiles based on machine learning methodologies. We will also establish a personalized epigenetic prediction model for allergy development and build the risk assessment platform for immunotoxicological reaction under tobacco smoke exposure. Finally, we will examine the causal relationship between epigenetic signatures and immunotoxicological reactions under an independent children's cohort.

DETAILED DESCRIPTION:
Teenager Smoking Reduction Trial (TSRT)

1. Study subjects

   TSRT is a solution-oriented trial aiming to evaluate the effectiveness of tobacco smoke reduction among teenagers. Eligible teenagers will fit the following criteria: (a) age between 12 and 16 years old; (b) have active smoke habits in past 6 months; (c) amount of smoke exceed 10 cigarettes per week. The subjects will be recruited from our previous database for schoolchildren. Telephone interview will be used to screen the eligibility for the teenagers. Recruitment will occur over 3-month period from 2011 April to June. The procedure for TSRT is showed in figure 2. In this plan, we will recruit at least 31 asthmatic children and 31 non-asthmatic children who have active smoke habits.
2. Data collection

A baseline data and at the 1-month and 2-month follow-up visits, the primary caregiver provided data by personal interview on parents reports. The demographic information in questionnaires included age, gender, level of education.

Teenagers will report the frequency of cigarette smoking by using a structured questionnaire. The definition of tobacco smoke exposure including: (a) ''Do you currently smoke?''-yes/no; (b) ''When did you begin to smoke regularly?''; (c) Smokers were also asked for the number of cigarettes they smoked on an average day. Nicotine dependence will be examined by using structure questionnaires from Fagerstrom model.

We will contact eligible teenagers individually to get informed consent before data collection. The effects of our teenager smoking reduction intervention program will be assessed by primary outcomes such as cotinine/creatinine ratio (CCR) and the status of tobacco smoke exposure from questionnaire. No matter which group the participant belongs to, intervention and usual control group, the secondary outcomes in all participants will be tested as follows:

1. Cytokines. We will test levels of interleukin 4, 5, 13 (IL-4, 5, 13), tumor necrosis factor-α (TNF-α), interferon-gamma (INF-γ) and toll-like receptors 2, 4, 9 (TLR-2, 4, 9).
2. Immunotoxicological reaction. We will determine levels of exhaled nitric oxide (eNO), serum eosinophil cationic protein (ECP) and absolute eosinophil count (AEC).
3. Oxidative stress markers. Levels of the markers 8-hydroxy-2-deoxyguanosine (8-OHdG), malondialdehyde (MDA) and F2-isoprostane (Iso-P) will be examined.

After first session is applied, all participants will be tested for primary outcomes and secondary outcomes at baseline, month 1 and month 3 of the intervention process. We can then compare the biomarkers before and after the intervention program.

ELIGIBILITY:
Inclusion Criteria:

(1) age between 12 and 16 years old; (2) Child had active smoking habit; and (3) have prior history of smoking habit.

Exclusion Criteria:

We will exclude children who do not fit in with the inclusion criteria.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in cotinine level at 3 months | 3 month
  Cotinine was the major proximate metabolite of nicotine,has been widely used as a biomarker of tobacco exposure. We will detect the urinary cotinine for children who had active smoking habit.
Change from Baseline in smoking status at 3 months | 3 months
  The smoking status for children will be measure by structure questionnaire.

SECONDARY OUTCOMES:
Change from Baseline in DNA methylation at 3 months | 3 months
Change from Baseline in immunological cytokine at 3 months | 3 months
Change from Baseline in miRNA expression at 3 months | 3 months
Change from Baseline in immunological function at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yungling Lee, Ph.D, Principal Investigator — National Taiwan University Hospital